CLINICAL TRIAL: NCT02160353
Title: Phase II Single-arm Study Evaluating Neo-adjuvant (Pre-radical Radiotherapy) Abiraterone Acetate (Plus Prednisolone) and Gonadotropin-Releasing Hormone (GnRH) Agonist in High Risk Localised Prostate Carcinoma
Brief Title: Neo-adjuvant Abiraterone Prostate Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE (ICORG) 13-23
Record Dates: First submitted 2014-06-04; First posted 2014-06-10 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: High Risk Localised Prostate Carcinoma
MeSH Terms: interventions — Abiraterone Acetate; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combined hormonal therapy (Experimental): Abiraterone acetate: 1000mg/day (four 250g tablets, orally once a day) for 126 days Prednisolone; 5mg/day (1 tablet orally once a day, concomitant to abiraterone acetate) for 126 days GnRh agonist for 4 injections (at 28 day intervals)
  Interventions: Drug: Abiraterone acetate, Prednisolone

INTERVENTIONS:
Drug: Abiraterone acetate, Prednisolone

SUMMARY:
The role of this study is to focus on the potential role of abiraterone acetate in treatment-naive patients newly diagnosed with high-risk localised prostate cancer requiring combined hormonal therapy and radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study related procedures
* Males aged 18 years or older
* ECOG performance status of less than or equal to 1
* Life expectancy of 10 years or more (using MSKCC nomogram)
* Pathological proven prostate carcinoma at intermediate to high risk of recurrence as defined by RTOG
* Clinically negative lymph nodes as established by imaging (pelvic CT / MRI), nodal sampling, or dissection within 60 days prior to registration, except patients with lymph nodes equivocal or questionable by imaging are eligible without biopsy if the nodes are less than or equal to 1.5cm; any node larger than this ion imaging will require negative biopsy for eligibility
* No evidence of bone metastases on bone scan within 60 days prior to registration. Equivocal bone scan findings are allowed if plain film x-rays are negative for metastasis.
* Clinical laboratory values during screening:

  * Haemoglobin greater than or equal to 10.0g/dl
  * Absolute neutrophil count (ANC) ≥ 1.8 × 10 to the power of 9/L
  * Platelets ≥ 100 × 10 to the power of 9/L
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 95 mmHg [Note: medically controlled hypertension is permitted]
* Prostate gland size measurable by trans-rectal ultrasound (TRUS) and at least greater than or equal to 30 cm cubed at baseline
* Patient is willing to use barrier-method of contraception along with another effective contraceptive method if engaged in sexual activity with a pregnant woman or a woman of child-bearing potential (until 1 week after completing treatment)

Exclusion Criteria:

* Prior treatment for prostate carcinoma, including prostatectomy; high intensity focused ultrasound or cryotherapy; hormonal manipulation (any modalities) including LHRH agonist, anti-androgen, or bilateral orchidectomy; prior or concomitant chemotherapy for prostate cancer; prior radiotherapy including brachytherapy to the region of study cancer; radical local treatment [Exception: Transuretheral Resection of the Prostate (TRUP) / TRUS is allowed]
* Use of urethral catheter
* History of cardiovascular disease; Uncontrolled hypertension [hypertension controlled by anti-hypertensive therapy is permitted], clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association Class III or IV heart failure, or Class II to IV heart failure of cardiac ejection fraction measurement of <50%
* Active or symptomatic viral hepatitis or chronic liver disease
* Major thoracic or abdominal surgery or significant traumatic injury within 4 weeks prior to registration, or planned surgery during study participation / within 4 weeks from end of treatment [Note: patients with planned surgical procedures to be conducted under local anaesthesia are not excluded from the study]
* Gastrointestinal disorder interfering with study drug absorption
* Active or uncontrolled disease that may require oral corticosteroid therapy
* Positive serology for hepatitis B surface antigen or hepatitis C antibody
* Known allergies, hypersensitivity or intolerance to abiraterone acetate, prednisolone, GnRH agonists or their excipients
* Contraindications to the use of prednisolone or GnRH agonists per local prescribing information
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study
* Any condition that, in the opinion of the investigator, would compromise the well-being of the patient or that could prevent, limit, or confound the protocol-specified assessments
* The patient has or had othe co-existing malignancies within the past 5 years, other than resected non-melanoma skin cancer
* Treatment with non-approved or investigational drug within 30 days before the first planned dose of study drug

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Clinical tumour response | 126 days
  To evaluate the clinical tumour response achieved by 126 days of neo-adjuvant combined treatment by abiraterone acetate, prednisolone and GnRH agonist in treatment of naive high-risk localised prostate carcinoma patients (prior to radical radiotherapy)
Biochemical response | 126 days
  To evaluate biochemical response achieved by 126 days of neo-adjuvant combined treatment by abiraterone acetate, prednisolone and GnRH agonist - in treatment naive high-risk localised prostate carcinoma patients (prior to radical radiotherapy)
Mean percentage reduction in prostate gland volume | 126 days
  To evaluate the mean percentage reduction in prostate gland volume achieved by 126 days of neo-adjuvant combined treatment by abiraterone acetate, prednisolone and GnRH agonist - in treatment naive high-risk localised prostate carcinoma patients (prior to radical radiotherapy)

SECONDARY OUTCOMES:
Testosterone level | 126 days
  To report the decrease in testosterone level

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Thirion, Dr, Principal Investigator — St Luke's Radiation Oncology Network, St Luke's Hospital
Locations (3):
- Ireland (3):
  - Cork University Hospital, Cork
  - St Luke's Hospital, Dublin
  - University Hospital Galway, Galway